CLINICAL TRIAL: NCT00386659
Title: A Randomized, Pilot Study on the Antiviral Activity and Immunological Effects of Lopinavir/Ritonavir vs. Efavirenz in Treatment-naïve HIV-Infected Patients With CD4 Cell Counts Below 100 Cells/mm3
Brief Title: Immune Reconstitution in naïve HIV Patients With CD4 <100 Cells/mL When Treated With Lopinavir or Efavirenz.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADVAN-Z-2
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2006-10

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; abacavir; Lopinavir; Ritonavir; efavirenz

INTERVENTIONS:
Drug: tenofovir + abacavir + lopinavir/ritonavir
Drug: tenofovir + abacavir + efavirenz

SUMMARY:
Pilot, randomized, parallel, open-label, controlled, clinical study evaluating virological response in plasma and extra-plasmatic compartments, together with the degree and kinetics of immune reconstitution in treatment-naïve patients with CD4 count below 100 cells/mL, when treated with tenofovir and abacavir together with lopinavir or efavirenz.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infection
* Antiretroviral-naive
* CD4 cell count below 100 cells/mm3

Exclusion Criteria:

* Pregnancy
* Current opportunistic infection requiring parenteral therapy
* Current malignancies requiring parenteral chemotherapy
* Any contraindication to the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60

PRIMARY OUTCOMES:
Proportion of patients with viral load below 20 copies/ml in plasma and lymphoid tissue at 12 months.

SECONDARY OUTCOMES:
Degree and kinetics of recovery of the immune system.
New CDC C events
Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Gatell, MD, Study Chair — Hospital Clinic of Barcelona
Locations (4):
- Spain (4):
  - Hospital de Sant Pau, Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - Hospital Clinic, Barcelona, Barcelona
  - CSU Bellvitge, L'Hospitalet de Llobregat, Barcelona